CLINICAL TRIAL: NCT06428513
Title: SHEBA-9466-22-RP-CTIL Health Coaching Telemedicine Program for Lung Transplant Candidates With End-stage Lung Disease: A Feasibility Study
Brief Title: Health Coaching Telemedicine Program for Lung Transplant Candidates With End-stage Lung Disease.
Acronym: HCTP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 9466-22-SMC
Record Dates: First submitted 2023-11-22; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2023-08

CONDITIONS: Copd; End Stage Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HCTP program (Experimental): Complete a HCTP program which includes 12 weekly one-on-one 30-minute tele-sessions through Zoom. Follow up will be for a year in total.
  Interventions: Behavioral: HCTP
- Control (No Intervention): Control group participants do not receive the intervention but will receive HCTP after the end of the study.

INTERVENTIONS:
Behavioral: HCTP — 10 weekly 1-on-1 30-minute tele-sessions via Zoom, delivered by a certified health coach. At baseline assessment including full medical history, medications, lifestyle practices, self-reported health status, psychosocial status, and other relevant information will be taken. At the first session, participants identify their health vision and 3-month health goals. At subsequent meetings, participants review their progress towards reaching the prior week's goals and identify goals for the next week. An individualized action plan will be formulated to help each participant achieve their goals. The action plan will focus on important lifestyle practices (physical activity/exercise training, correct nutrition, weight management, tobacco cessation, and stress management. Patients can request further health care advice felt necessary for their progress, and will be referred to health care professionals in the rehabilitation hospital that provide care for lung transplantation candidates.
  Other Names: Health coaching telemedicine program
  Arms: HCTP program

SUMMARY:
Lung transplantation has become standard of care for selected patients with end stage pulmonary disease. While on the lung transplantation waiting list, patient health, emotional wellbeing and quality of life can deteriorate. By improving or changing patient physical activity, healthy nutrition, tobacco cessation, patient preparation for lung transplantation can be optimized, risk of complications can be reduced, and outcomes post transplantation can be improved.

The potential of health coaching to improve health outcomes has been demonstrated in several chronic diseases such as type 2 diabetes mellitus, congestive heart failure, and rheumatoid arthritis. In addition, health coaching was proven effective through telemedicine.

No studies so far have addressed the potential effect of a pre-transplant health coaching program on existing medical conditions, transplant rates and post-transplant outcomes. Investigators hypothesized that health coaching can improve health outcomes and survival of lung transplantation candidates by supporting and growing patients' capacity to cope with the demands of their end stage pulmonary disease.

DETAILED DESCRIPTION:
SCIENTIFIC BACKGROUND Lung transplantation has become an established standard of care for selected patients with end stage pulmonary disease. Candidate selection begins with a referral from the non-transplant pulmonologist and if deemed suitable, begins an evaluation process that determines eligibility for transplantation. Candidates who meet all requirements are listed for transplantation. While on the waiting list, physical activity, healthy nutrition, tobacco cessation, and a few other health behaviors are essential to maintain candidacy. In addition to the physical limitations imposed by end-stage lung disease, transplant candidates face a range of psychosocial issues relating to changes in functional capacity, including social roles, relationships, perceptions of self, and life plans and goals. Efforts targeted at these domains may improve quality of life, optimize patient preparation for transplantation, reduce the risk of complications, and improve outcomes.

Health coaching has emerged as a widely adopted intervention that may help individuals with chronic conditions adopting health behaviors that improve quality of life, health, and emotional wellbeing. It is a patient-centered approach wherein the individual and coach work together through active health education processes and motivational interviewing to set goals that improve health outcomes. The potential of health coaching to improve health outcomes has been demonstrated in several chronic diseases such as type 2 diabetes mellitus, congestive heart failure, and rheumatoid arthritis. In addition, health coaching was proven effective through telemedicine; and recently, it has developed national standards and accreditations in the US. Therefore, health coaching was selected as our telemedicine approach, and a novel health coaching telemedicine program (HCTP) was developed at Sheba Medical Center for lung transplantation candidate.

No studies so far have addressed the potential effect of pre-transplant health coaching program on existing medical conditions, transplant rates and post-transplant outcomes. Investigators hypothesized that health coaching can improve health outcomes and survival of lung transplantation candidates by supporting and growing patients' capacity to cope with the demands of their end stage pulmonary disease.

SPECIFIC AIMS Specific Aim 1: To assess whether HCTP is feasible among participants with end stage lung disease who are candidate for lung transplantation.

Specific Aim 2: To collect data on the impact of a HCTP on health-related quality of life, lung functions, functional capacity, cardiometabolic parameters (e.g., weight, lipid profile, fasting glucose), and hospital services utilization of participants with end stage lung disease who are candidate for lung transplantation Specific Aim 3: To collect data on experience and capacity to cope with the demands of the illness of participants with end stage lung disease who are candidate for lung transplantation.

STUDY DESIGN Detailed Plan of the Study The health coaching tele-medicine program study is a randomized controlled feasibility trial in which study participants are randomly assigned into either a study group or a control group.

Source of participants and recruitment methods: This study is a collaboration between the lung transplant program and the center of lifestyle medicine, within Sheba's cardiometabolic prevention center, a unique center in Israeli health care services that promote innovative lifestyle interventions. Our target population is 56 adults with end stage lung disease who refer to The Sheba Medical Center lung transplantation program for evaluation; over a period of 12 months.

METHODS:

This study is expected to be ongoing for 24 months but conducted for each subject in a 12-month timeframe. Data collection time points every quarter for 12 months.

Assessment include:

* Health related quality of life (HRQL)
* Lung functions tests
* Hospital services usage: will be evaluate using the hospital medical record. These services include health professional services in the rehabilitation hospital.
* Health behaviors: Nutritional intake will be evaluated by a 4-day food record.
* Physical activity questionnaire.
* Cardiometabolic outcomes
* Qualitative data: Investigators also expect to deepen our understanding about participants' experience in the program and their capacity to cope with the demands of their illness through the study's qualitative component. Qualitative data will be included in analyses for both participants who completed the intervention and participants who dropout.

Information regarding demographics, medications, other health behaviors (e.g., smoking status, physical activity status), and use of other nutritional education resources during the program (e.g., dietitian and physician visits, apps) will be extracted from the medical record.

PROCEDURE INTERVENTION: Both the intervention and control groups will receive the standard care for lung transplantation candidates. In addition for:

Study group participants - study group participants will complete a HCTP program which includes 12 weekly one-on-one 30-minute tele-sessions through Zoom, delivered by a credential health coach (health care professional who also completed a health coaching certification). Prior to the beginning of the program participant will complete intake assessment that will include past and current medical history, medications, current lifestyle practices, self-reported health status, psychosocial status, and other relevant information. At the first session, participants identify their health vision and 3-month health goals. During each subsequent meeting, participants will review their progress towards reaching the prior week's goals and identify goals for the coming week, using a self-discovery process facilitated by the health coach. Based on the initial assessment individualized action plan will be formulated to help each participant achieve his/her goals. The action plan will focus on important lifestyle practices (especially physical activity/exercise training, correct nutrition, weight management, tobacco cessation, and stress management. Based on their interaction with the participant and/or input from the participant's physician or other health care providers, health coaches will revise goals and action plans. When patients detect the need for health care advice that is necessary for their progress, s/he will be referred to health care professionals in the rehabilitation hospital that provide care for lung transplantation candidate.

2. Control group: Control group participants will receive HCTP after the end of the study.

Statistical methods: Patients will be randomized 1:1 between the 2 study arms. Investigators will use block randomization stratified by site. Power calculation indicates that 28 participants (14/ group) are required in each of the intervention groups in order to estimate a retention rate of 80% with 10% precision and 80% confidence. Every effort will be made to minimize dropouts, and further to follow-up with participants who do not complete the program to obtain measurements of study outcomes. In the event of missing data, the impact will be assessed and addressed, if necessary, according to current best practices. Demographic and other baseline characteristics as well as feasibility outcomes will be summarized using means and standard deviations for normally distributed variables, medians and interquartile ranges for non-normally distributed variables, and frequencies for count or dichotomous variables. For all outcomes and to address exploratory hypotheses. P-values and 95% confidence intervals will be presented for all effects of interest.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with end stage lung disease assessed suitable for lung transplantation.
* Able and willing to watch online instructional videos.

Exclusion Criteria:

* Unwilling or unable to provide consent
* Uncooperative or combative
* Unable to use / connect to video conferencing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-11-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility outcomes | Every quarter for one year
  Retention of participants in the program/research. Calculated as a percentage of participants completing all visits of the intervention.
Participant adherence | Every quarter for one year
  Participant percentage that adhered to the intervention. Calculated as a percentage of the intervention.
Forced expiratory volume in one second (FEV1) and Forced vital capacity (FVC) ratio: FEV1/FVC Ratio | Every quarter for one year
  FEV1/FVC ratio expressed as a percentage. The lower the percentage, the more severe the lung condition.
  Predictive (normal) values are equal to or greater than 70%. Abnormal values are graded:
  Mild: 60-69% Moderate: 50-59% Severe: Under 50%
Total lung capacity (TLC) | Every quarter for one year
  Total lung capacity (TLC), recorded in Liters (L)
Diffusing capacity of the lungs for carbon monoxide (DLCO) | Every quarter for one year
  Changes in DLCO test from the baseline used to determine progression or regression of disease.
  DLCO (also known as Transfer factor for carbon monoxide (TLCO)) Units ml/min/mmHg/L. Initial and final Carbon monoxide (CO) concentration, in mmol CO, and breath-holding time in minutes, are used to calculate DLCO
  Severity and classification of DLCO reduction:
  Normal DLCO: >75% of predicted, up to 140% Mild: 60% to LLN (lower limit of normal) Moderate: 40% to 60% Severe: <40%
Functional lung capacity using six-minute walk test (6MWT) | Every six months for one year
  To assess a patient's functional status / to track functional change resulting from disease progression or therapeutic intervention.
  The higher a patient's score, the better their lung capacity. A low score correlates with lower function.
  Calculation measurements: weight in kilograms, height in centimetres, age of patient in years, distance walked meters.
  Calculation
  MEN:
  6MWD = (7.57 × height) - (5.02 × age) - (1.76 × weight) - 309
  WOMEN:
  6MWD = (2.11 × height) - (2.29 × weight) - (5.78 × age) + 667
  Heart rate and oxygen saturation will also be measured separately but included to provide an assessment of functional status.
Oxygen saturation | Every six months for one year
  Oxygen saturation, measured as a percentage. Taken at rest and breathing room air, and during taken during exercise test.
  This is used as part of Functional lung capacity using six-minute walk test (6MWT) to assess functional capacity.
Heart Rate | Every six months for one year
  Heart Rate measured as a beats per minute. Taken at rest and breathing room air, and during taken during exercise test.
  This is used as part of Functional lung capacity using six-minute walk test (6MWT) to assess functional capacity.
Physical activity variable | Every quarter for one year
  Physical activity will be measured by the international physical activity questionnaire. A change in physical activity
  Scoring a HIGH level of physical activity on the IPAQ means the participant's physical activity levels equate to approximately one hour of activity per day or more at least a moderate intensity activity level.
  Scoring a MODERATE level of physical activity on the IPAQ means the participant is doing some activity more than likely equivalent to half an hour of at least moderate intensity physical activity on most days.
  Scoring a LOW level of physical activity on the IPAQ means that the participant is not meeting any of the criteria for either MODERATE of HIGH levels of physical activity.
Behavioural and nutritional evaluation | Every quarter for one year
  • Health behaviours: Nutritional intake will be evaluated by a 4-day food record in which subjects document and report their food consumption. Intake will be analyzed for its caloric content, nutritional values and group classifications and its Mediterranean index.
Patient functioning and quality of life | Every quarter for one year
  Evaluated using the St. George's respiratory questionnaire. Disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease.Scores range from 0 to 100, with higher scores indicating more limitations.

SECONDARY OUTCOMES:
Body mass index (BMI) | Every quarter for one year
  Height (cm) and weight (kg) will be combined to report BMI in kg/m^2
Glucose control - glycated hemoglobin HbA1c | Every quarter for one year
  Hemoglobin A1c (glycated hemoglobin), HbA1c measured as percentage (%)
  Changes in measurements between visits over time will be analysed.
Blood lipid profile | Every quarter for one year
  Includes total cholesterol, HDL-cholesterol, LDL-cholesterol, non-HDL cholesterol and triglycerides. Measured in milligrams (mg) of cholesterol per deciliter (dL) of blood (mg/dl)
  Changes in measurements between visits over time will be analysed.
Cardio-metabolic evaluation | Every quarter for one year
  Cardio-metabolic outcomes: (2) blood pressure systolic and diastolic
  Changes in measurements between visits over time will be analysed.
Rate of hospital service usage | One year
  Changes in the number of hospital services / engagements used i.e., physiotherapist, social worker, nutritionist, hospitalizations, and emergency room admissions engagements per month.
Participant perception of the program | Month 0
  Qualitative data: To deepen our understanding about subjects' experience in the program and their capacity to cope with the demands of their illness through the study's qualitative component. Qualitative data will be included in analyses for both subjects who completed the intervention and subjects who dropout.Baseline/Visit 1 - a questionnaire with open questions to fill out about the subject's challenges and expectations before the program starts (both intervention and control group).
Behavioural and psychosocial outcome | Month 3
  Qualitative data Visit 2 - a questionnaire with open retrospective questions to fill out about the subject's experience at the HCTP (Intervention group only)
Participant evaluation | Month 6
  Qualitative data Visit 3 - a follow-up interview to sum up the subject's experience

CONTACTS AND LOCATIONS:
Overall Officials: Rani Polak, PhD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No